CLINICAL TRIAL: NCT02364024
Title: Biomarker Validation Study of Linear Quantification of CD3 Positive Cells in Localized Colorectal Carcinomas, Based on the Cohort of Patient Included in PETACC8 International Phase III Trial (NCT00265811)
Brief Title: Validation Study of Linear Quantification of CD3+ Cells in Localized Colorectal Carcinomas
Acronym: CD3-OncoQuant
Status: Completed | Type: Observational
Sponsor: Federation Francophone de Cancerologie Digestive (Other)
Responsible Party: Sponsor
Other Study IDs: PETACC8-BIO1
Record Dates: First submitted 2015-02-10; First posted 2015-02-16 (Estimated); Last update posted 2018-07-06 (Actual); Status verified 2018-07

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Colon and rectum carcinoma; Immune response; Biomarker; Prognosis
MeSH Terms: conditions — Colorectal Neoplasms; Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissues: colorectal carcinoma and adjacent non-tumor tissues are collected in formalin fixed paraffin embedded blocks.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Arm A: Patients with no or low immune response (score 1 or 2) with linear quantification of CD3+ cells
- Arm B: Patients with high immune response (score 3 or 4) with linear quantification of CD3+ cells

SUMMARY:
The purpose of this study is to confirm that linear quantification of CD3+ cells is a prognostic biomarker in localized colorectal carcinomas.

DETAILED DESCRIPTION:
Adult patients of both gender who have underwent surgical resection of stage III colorectal carcinoma and randomised to receive a chemotherapy FOLFOX or FOLFOX + Cetuximab in the PETACC8 trial.

ELIGIBILITY:
Inclusion Criteria:

* Patient included in PETACC08 study
* Signed informed consent for translational study
* FFPE tumor sample available for CD3 staining

Exclusion Criteria:

- Patient who have withdrawn their consent for PETACC08 and/or for PETACC08 translational study

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patient of both gender who have underwent surgical resection of stage III colorectal carcinoma
Sampling Method: Probability Sample
Enrollment: 856 (Actual)
Dates: Start 2005-11; Primary Completion 2009-05 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Time to Recurrence (TTR) | 2 years
  TTR is defined by the time between randomisation and the first event occured (Local or metastatic recurrence or death due to disease recurrence) whichever occured first or last follow-up ( Last news for patients without event (censored data))

SECONDARY OUTCOMES:
Overall Survival (OS) | until death
  Overall survival is defined as the time from randomization to death any cause or last follow-up news (censored data).
Disease-Free Survival (DFS) | 2 years
  DFS is defined by the time between randomisation and the first event occured (Local or metastatic recurrence or second cancer or death (all causes)) whichever occured first or last follow-up ( Last news for patients without event (censored data))

CONTACTS AND LOCATIONS:
Overall Officials: Emile Jean-François, Pr, Study Director — Fédération Fancophone de Cancérologie Digestive

REFERENCES:
- [Background] Taieb J, Tabernero J, Mini E, Subtil F, Folprecht G, Van Laethem JL, Thaler J, Bridgewater J, Petersen LN, Blons H, Collette L, Van Cutsem E, Rougier P, Salazar R, Bedenne L, Emile JF, Laurent-Puig P, Lepage C; PETACC-8 Study Investigators. Oxaliplatin, fluorouracil, and leucovorin with or without cetuximab in patients with resected stage III colon cancer (PETACC-8): an open-label, randomised phase 3 trial. Lancet Oncol. 2014 Jul;15(8):862-73. doi: 10.1016/S1470-2045(14)70227-X. Epub 2014 Jun 11. PMID 24928083
- [Result] Emile JF, Julie C, Le Malicot K, Lepage C, Tabernero J, Mini E, Folprecht G, Van Laethem JL, Dimet S, Boulagnon-Rombi C, Allard MA, Penault-Llorca F, Bennouna J, Laurent-Puig P, Taieb J; PETACC8 Study Investigators; Austrian Breast and Colorectal cancer Study Group (ABCSG); Belgian Group of Digestive Oncology (BGDO); Lone Norgard Petersen; Federation Francophone de Cancerologie Digestive (FFCD); Federation Nationale des Centres de Lutte Contre le Cancer (UNICANCER); Federation Nationale des Centres de Lutte Contre le Cancer Association Europeenne de Recherche en Oncologie (AERO); Arbeitsgemeinschaft Internistische Onkologie (AIO); Gruppo Italiano per lo Studio dei Carcinomi dell'Apparato Digerente (GISCAD); Gruppo Oncologico dell'Italia Meridionale (GOIM); Istituto Oncologico Romagnolo (IOR); Gruppo Cooperativo Chirurgico Italiano (GOCCI); Gruppo Oncologico Nord Ovest (GONO); Gruppo Oncologico Italiano di Ricerca Clinica (GOIRC); Gruppo Cooperativo do Cancro Digestivo da Associacao Portuguesa de Investigacao Oncologica (GCCD, APIO); Grupo Espanol para el Tratamiento de los Tumores Digestivos (TTD); John Allen Bridgewater. Prospective validation of a lymphocyte infiltration prognostic test in stage III colon cancer patients treated with adjuvant FOLFOX. Eur J Cancer. 2017 Sep;82:16-24. doi: 10.1016/j.ejca.2017.04.025. Epub 2017 Jun 23. PMID 28651158